CLINICAL TRIAL: NCT00783354
Title: A Pilot, Multicenter, Double-blind Randomized Study for Comparison of Aerius® "Continuous Treatment" Versus Aerius® "PRN Regimen" on Chronic Idiopathic Urticaria Patient Quality of Life
Brief Title: A Comparison of Aerius Continuous Treatment Versus Aerius PRN for Chronic Idiopathic Urticaria (Study P03147)
Acronym: ATTITUD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P03147
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Urticaria; Chronic Idiopathic Urticaria
MeSH Terms: conditions — Urticaria; Chronic Urticaria | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Treatment (Active Comparator)
  Interventions: Drug: desloratadine
- PRN regimen (Experimental)
  Interventions: Drug: desloratadine

INTERVENTIONS:
Drug: desloratadine — Patients received desloratadine 5 mg daily, given as one tablet in the evening, and were asked to take one tablet of "rescue medication" (Placebo) in case of symptoms for 2 months.
  Other Names: Aerius; SCH 34117
  Arms: Continuous Treatment
Drug: desloratadine — Patients received Placebo daily, given as one tablet in the evening, and were asked to take one tablet of "rescue medication" (desloratadine 5 mg) in case of symptoms for 2 months.
  Other Names: Aerius; SCH 34117
  Arms: PRN regimen

SUMMARY:
This double-blind pilot study was conducted to establish the best way of using desloratadine treatment to protect quality of life of chronic idiopathic urticaria (CIU) patients, after an initial 4-weeks of daily treatment: prolonging systematic daily treatment or as needed (PRN; in the case of symptoms).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects must be >= 18 years of age
* Women of childbearing potential must have a negative urine pregnancy test at Visit 1 (Day 1) and must be using an acceptable method of birth control during the study.
* Subjects must be in general good health; ie, they must be free of any clinically significant disease (other than CIU) that would interfere with study evaluations.
* Subjects must understand and be able to adhere to visit schedules, and agree to complete the questionnaires and a diary.
* Subjects must have at least a 6-week history of CIU (pruritus and hives) prior to Visit 1.

Exclusion Criteria:

* Women who are pregnant or nursing.
* Subjects who used any investigational drug in the last 30 days prior to Visit 1
* Subjects with asthma requiring chronic use of inhaled or systemic corticosteroids.
* Subjects who have been treated with any investigational antibodies for asthma or allergic rhinitis in the 90 days prior to Baseline.
* Subjects who have been treated with intra-muscular or intra-articular corticosteroids in the 90 days prior to Baseline.
* Subjects with urticaria that is primarily due to physical urticaria or other known etiology, except dermographism.
* Subjects treated by immunosuppressive drugs.
* Subjects who have been hospitalized (including an emergency department visit) because of deterioration in their CIU within 3 months prior to Visit 1.
* Subjects with a history of hypersensitivity to desloratadine or any of its excipients.
* Subjects previously randomized into this study.
* Subjects who have any clinically significant metabolic, cardiovascular, immunological, neurological, hematological, gastrointestinal, cerebrovascular, or respiratory disease, or any other disorder which, in the judgment of the investigator, may interfere with the study evaluations or affect subject safety.
* Subjects with a history of psychosis, antagonistic personality, poor motivation, hypochondriasis, or any other emotional or intellectual problems that are likely to limit the validity of consent to participate in the study.
* Subjects with a history of noncompliance with medications or treatment protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2003-04-01 (Actual); Primary Completion 2004-02-01 (Actual); Study Completion 2004-04-01 (Actual)

PRIMARY OUTCOMES:
Changes from Visit 2 to Visit 4 of Vq-derm questionnaire score and DLQI quality of life score. | 2 months

SECONDARY OUTCOMES:
Estimation of disease free period after 3 months of daily treatment. | 2 months
Average usage of rescue medication | 2 months
Change from Visit 2 in pruritus symptom score assessed by the patient. | 2 months
% of patients free of symptoms 2 months after Visit 4 | 2 months
Changes from Visit 2 of overall conditions of CIU | 2 months
Discontinuation due to treatment failure | 2 months
Investigator's assessment of response to therapy | 2 months
Quality of disease control | 2 months
Average consumption of treatment between Visit 2 and Visit 5 | 4 months

REFERENCES:
- [Result] Grob JJ, Auquier P, Dreyfus I, Ortonne JP. How to prescribe antihistamines for chronic idiopathic urticaria: desloratadine daily vs PRN and quality of life. Allergy. 2009 Apr;64(4):605-12. doi: 10.1111/j.1398-9995.2008.01913.x. Epub 2008 Dec 30. PMID 19133920